CLINICAL TRIAL: NCT03706872
Title: Efficacy of an App for Monitoring Physical Activity and Weight of Obese Pregnant Women
Brief Title: Efficacy of an App for Monitoring Physical Activity and Weight of Obese Pregnant Women (Pas&Pes)
Acronym: Pas&Pes
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Women's confinement for COVID-19 pandemic and changes on prenatal care.
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Elena Gonzalez-Plaza, Midwife, Hospital Clinic of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HCB2017/0756
Record Dates: First submitted 2018-10-10; First posted 2018-10-16 (Actual); Last update posted 2020-05-18 (Actual); Status verified 2020-05

CONDITIONS: Obese Pregnant Women
Keywords: pregnant women; obesity; Mobile Applications; weight gain; physical activity
MeSH Terms: conditions — Obesity; Weight Gain; Motor Activity

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial with 2 arms of intervention
Who Masked: Care Provider
Masking Description: Care provider will not know the arm of randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The provision of an App for monitoring physical activity and weight with a smart watch and the administration of virtual advice through messages with mobile phone and the midwife's feedback, as well as the provision of usual prenatal care.
  Interventions: Other: Intervention group
- Control Group (No Intervention): Provision of usual prenatal care

INTERVENTIONS:
Other: Intervention group — The provision of an App for monitoring physical activity and weight with a smart watch and the administration of virtual advice through messages with mobile phone and the midwife's feedback, as well as the provision of usual prenatal care
  Arms: Intervention group

SUMMARY:
This study evaluate the efficacy of an App for monitoring the physical activity and weight with a smart watch and the provision of virtual advice through messages with a mobile phone in obese pregnant women in the second trimester.

Half of the women will be randomized at the intervention group (App + smart watch) and the other half, to the control group who will receive the usual prenatal care.

DETAILED DESCRIPTION:
Randomized controlled trial among obese women. These women will be randomized in two groups in order to evaluate an improvement in several outcomes thanks to different strategies:

Intervention group (IG). An App for monitoring physical activity and weight with a smart watch and the administration of virtual advice through messages with mobile phone and the midwife's feedback, as well as the provision of usual prenatal care.

Control group. Pregnant women will receive the usual prenatal care. Main hypothesis: In the intervention group pregnant women will improve the weight gain adjusted to the preconception BMI, during pregnanacy, with respect to the pregnant women of the control group.

Secondary hypothesis. In the intervention group pregnant women will improve the physical activity.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with BMI ≥ 30 Kg / m2 preconceptional
* Speak Spanish fluently
* Viable singleton non-malformed fetus
* 12-18 weeks of gestation
* Users of Android or Iphone smart mobile phone with internet connection

Exclusion Criteria:

* Pregnant women users of a physical activity and weight monitoring App
* Pregnant women with Type I or II Diabetes Mellitus
* Pregnant Women with psychiatric disorders
* Pregnant women with thyroid disorders
* Women with chronic hypertension
* Pregnant women who for some reason have contraindicated the performance of exercise or mobility problems that make it impossible to walk in a moderate way.
* Pregnant women who do not accept to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Gestational weight gain | 36 weeks
  Compare gestational weight gain dring pregnancy in both groups.
Physical activity | 36 weeks
  METS/minutes/week by the "IPAQ Scale" short version

SECONDARY OUTCOMES:
Gestational complications | 36 weeks
  Prevalence of preeclampsia, gestational diabetes.
Intrapartum complications | Labor
  Labor inductions and type of labor
perinatal complications | birth
  Prevalence of prematurity, macrosomia

OTHER OUTCOMES:
App usability | 36 weeks
  To describe the App usability using "System Usability Scale" in pregnant women of the experimental group
Eating habits | 36 weeks
  Compare eating habits in both groups with "dietary habits questionaire for the overweight and obese"

CONTACTS AND LOCATIONS:
Overall Officials: Elena González-Plaza, Midwife, Principal Investigator — Clinic Hospital of Barcelona; Gloria Seguranyes, PhD, Study Director — University of Barcelona; Jordi Bellart, PhD, Study Director — Clinic Hospital of Barcelona
Locations (1):
- Elena González-Plaza, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonzalez-Plaza E, Bellart J, Arranz A, Lujan-Barroso L, Crespo Mirasol E, Seguranyes G. Effectiveness of a Step Counter Smartband and Midwife Counseling Intervention on Gestational Weight Gain and Physical Activity in Pregnant Women With Obesity (Pas and Pes Study): Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Feb 15;10(2):e28886. doi: 10.2196/28886. PMID 35166684